CLINICAL TRIAL: NCT05471284
Title: A Multimethod Evaluation of Tobacco Treatment Trial Recruitment Messages for Current Smokers Recently Diagnosed With Cancer: Pilot Factorial Randomized Controlled Trial
Brief Title: Recruitment Messages for Current Smokers Recently Diagnosed With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Tufts University (Other); Massachusetts General Hospital (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018P002035
Record Dates: First submitted 2022-07-13; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Tobacco Smoking; Health Behavior
Keywords: Cancer; Digital outreach; Multimethod randomized trial; Factorial Design; Message Frames; Tobacco use; Smoker enrollment rates
MeSH Terms: conditions — Tobacco Smoking; Health Behavior; Neoplasms; Tobacco Use | interventions — Costs and Cost Analysis; Gain of Function Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Control (Sham Comparator): The control condition was a kernel message that included study information present in all conditions but did not include any of the message factors.
  Interventions: Behavioral: Control
- Proximal x Cost x Loss (Experimental): Message frame: proximal threats of smoking, cost of continued smoking, and loss of not participating in a tobacco treatment trial.
  Interventions: Behavioral: Proximal; Behavioral: Cost; Behavioral: Loss
- Proximal x Cost x Gain (Experimental): Message frame: proximal threats of smoking, cost of continued smoking, and gain of participating in a tobacco treatment trial.
  Interventions: Behavioral: Proximal; Behavioral: Cost; Behavioral: Gain
- Proximal x Benefit x Gain (Experimental): Message frame: proximal threats of smoking, benefits of quitting, and gain of participating in a tobacco treatment trial.
  Interventions: Behavioral: Proximal; Behavioral: Benefit; Behavioral: Gain
- Proximal x Benefit x Loss (Experimental): Message frame: proximal threats of smoking, benefits of quitting, and loss of not participating in a tobacco treatment trial.
  Interventions: Behavioral: Proximal; Behavioral: Benefit; Behavioral: Loss
- Distal x Cost x Gain (Experimental): Message frame: distal threats of smoking, cost of continued smoking, and gain of participating in a tobacco treatment trial.
  Interventions: Behavioral: Distal; Behavioral: Cost; Behavioral: Gain
- Distal x Cost x Loss (Experimental): Message frame: distal threats of smoking, cost of continued smoking, and loss of not participating in a tobacco treatment trial.
  Interventions: Behavioral: Distal; Behavioral: Cost; Behavioral: Loss
- Distal x Benefit x Loss (Experimental): Message frame: distal threats of smoking, benefits of quitting, and loss of not participating in a tobacco treatment trial.
  Interventions: Behavioral: Distal; Behavioral: Benefit; Behavioral: Loss
- Distal x Benefit x Gain (Experimental): Message frame: distal threats of smoking, benefits of quitting, and gain of participating in a tobacco treatment trial.
  Interventions: Behavioral: Distal; Behavioral: Benefit; Behavioral: Gain

INTERVENTIONS:
Behavioral: Proximal — The first factor tested framing of the near, proximal threat of continued smoking.
  Arms: Proximal x Benefit x Gain; Proximal x Benefit x Loss; Proximal x Cost x Gain; Proximal x Cost x Loss
Behavioral: Distal — The first factor tested framing of the long-term, distal threat of continued smoking.
  Arms: Distal x Benefit x Gain; Distal x Benefit x Loss; Distal x Cost x Gain; Distal x Cost x Loss
Behavioral: Cost — Cost framework measures the response efficacy to quitting smoking by displaying costs of continued smoking.
  Arms: Distal x Cost x Gain; Distal x Cost x Loss; Proximal x Cost x Gain; Proximal x Cost x Loss
Behavioral: Benefit — Benefit framework measures the response efficacy to quitting smoking by displaying benefits of quitting.
  Arms: Distal x Benefit x Gain; Distal x Benefit x Loss; Proximal x Benefit x Gain; Proximal x Benefit x Loss
Behavioral: Loss — The third factor tested framing of the response efficacy of participating in a cessation study by utilizing loss of not participating in a smoking cessation.
  Arms: Distal x Benefit x Loss; Distal x Cost x Loss; Proximal x Benefit x Loss; Proximal x Cost x Loss
Behavioral: Gain — The third factor tested framing of the response efficacy of participating in a cessation study by utilizing gain of participating in a smoking cessation.
  Arms: Distal x Benefit x Gain; Distal x Cost x Gain; Proximal x Benefit x Gain; Proximal x Cost x Gain
Behavioral: Control — Does not include any of the three message factors.
  Arms: Control

SUMMARY:
The objective of this study was to conduct a pilot factorial randomized trial to identify the message frames that are most effective in promoting participation in a tobacco treatment trial for current smokers recently diagnosed with cancer. To do so, we used a multimethod approach to evaluate 3 different message frames across evaluation, effectiveness, and outcome measures. We combine findings from a message design experiment with textual analytic software to provide a holistic understanding of how message frames may or may not differentially affect tobacco treatment trial participation within the context of a cancer diagnosis.

DETAILED DESCRIPTION:
Background: A cancer diagnosis can catalyze motivation to quit smoking. Tobacco treatment trials offer cessation resources but have low accrual rates. Digital outreach may improve accrual, but knowledge of how best to recruit smokers with recent diagnoses is limited.

Objective: This study aims to identify the message frames that were most effective in promoting intent to talk to a physician about participating in a tobacco treatment trial for smokers recently diagnosed with cancer.

Methods: From February to April 2019, current smokers diagnosed within the past 24 months were recruited from a national web-based panel for a multimethod pilot randomized trial (N=99). Participants were randomized to a 2×3 plus control factorial design that tested 3 unique message frames: proximal versus distal threats of smoking, costs of continued smoking versus benefits of quitting, and gains of participating versus losses of not participating in a tobacco treatment trial.

ELIGIBILITY:
Inclusion Criteria:

* Speak and understand English
* A recent cancer diagnosis (within the past 24 months)
* 18 years or older
* Report any cigarette use within the past 30 days

Exclusion Criteria:

* Do not speak or understand English
* Have not been diagnosed with cancer within the past 24 months
* Below the age of 18
* Does not report any cigarette use within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Difference in intent to talk to a physician about participating in a smoking cessation study between factors. | Within 30 minutes
  The main effect within each message factor level was examined using ANOVA and compared with the control condition.

SECONDARY OUTCOMES:
Predictors of intent to talk to a physician about participating in a smoking cessation study. | Within 30 minutes
  Other message evaluation and effectiveness measures were collected and explored in a multivariable model predicting intent to talk to a physician.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Neil, Ph.D., Principal Investigator — TSET Health Promotion Research Center
Locations (1):
- Jordan Neil, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neil JM, Senecal C, Ballini L, Chang Y, Goshe B, Flores E, Ostroff JS, Park ER. A Multimethod Evaluation of Tobacco Treatment Trial Recruitment Messages for Current Smokers Recently Diagnosed With Cancer: Pilot Factorial Randomized Controlled Trial. JMIR Cancer. 2022 Aug 24;8(3):e37526. doi: 10.2196/37526. PMID 36001378

DOCUMENTS (2):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT05471284/Prot_000.pdf
  • Informed Consent Form (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT05471284/ICF_001.pdf